CLINICAL TRIAL: NCT00032175
Title: A Phase III Multicenter Randomized Clinical Trial Comparing Gemcitabine Alone Or In Combination With Capecitabine For The Treatment Of Patients With Advanced Pancreatic Cancer
Brief Title: Gemcitabine With or Without Capecitabine in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CRUK-GEM-CAP; CDR0000069263 (Registry Identifier: PDQ (Physician Data Query)); EU-20116; ISRCTN11513444
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; duct cell adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Gemcitabine

INTERVENTIONS:
Drug: capecitabine
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if gemcitabine is more effective with or without capecitabine in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of gemcitabine with or without capecitabine in treating patients who have locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 1-year survival rate of patients with locally advanced or metastatic pancreatic cancer treated with gemcitabine with or without capecitabine.
* Compare the median and 2-year survival rates and the objective response rates of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is an randomized, open-label, multicenter study. Patients are stratified according to disease stage (locally advanced vs metastatic) and performance status (0 and 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43 during the first course. After a 1-week rest period, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Subsequent courses repeat every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 3 months for 1 year, and then annually thereafter.

Patients are followed every 3 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 508 patients (254 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed ductal adenocarcinoma of the pancreas

  * Locally advanced or metastatic disease not amenable to curative surgical resection
  * Macroscopic residual disease after prior resection with histological confirmation is allowed
* Unidimensionally measurable disease
* No intracerebral metastases or meningeal carcinomatosis

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* WHO 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC greater than 3,000/mm3
* Neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 2 mg/dL

Renal:

* Creatinine less than 2 mg/dL
* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No uncontrolled angina pectoris

Other:

* No other prior malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other concurrent uncontrolled medical condition
* No other medical or psychiatric condition that would preclude study
* No known hypersensitivity to fluorouracil
* No dihydropyrimidine dehydrogenase deficiency
* No known malabsorption syndromes
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy (including preoperative or adjuvant) for this disease
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy (including preoperative or adjuvant) for this disease

Surgery:

* See Disease Characteristics

Other:

* No prior investigational drugs (including preoperative or adjuvant) for this disease
* No other concurrent investigational drugs
* No concurrent dipyridamole or allopurinol
* No concurrent sorivudine or sorivudine analogs (e.g., brivudine) (capecitabine arm only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2002-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Survival at 1 year

SECONDARY OUTCOMES:
Quality of life
Median survival rate
Survival rate at 2 years
Toxicity
Objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Emily Owen — Cancer Research UK
Locations (30):
- United Kingdom (30):
  - Royal United Hospital, Bath, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - Cancer Research UK Liverpool Cancer Trials Unit, Liverpool, England
  - Royal Liverpool University Hospital, Liverpool, England
  - St. Thomas' Hospital, London, England
  - Christie Hospital NHS Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - James Cook University Hospital at South Tees Hospitals NHS Trust, Middlesbrough, Cleveland, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Derriford Hospital, Plymouth, England
  - Poole Hospital NHS Trust, Poole Dorset, England
  - Whiston Hospital, Prescot Merseyside, England
  - Royal Preston Hospital, Preston, England
  - Salisbury District Hospital, Salisbury, England
  - Royal South Hants Hospital, Southampton, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Warrington Hospital NHS Trust, Warrington, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Singleton Hospital of the Swansea NHS Trust, Swansea, Wales

REFERENCES:
- [Result] Cunningham D, Chau I, Stocken DD, Valle JW, Smith D, Steward W, Harper PG, Dunn J, Tudur-Smith C, West J, Falk S, Crellin A, Adab F, Thompson J, Leonard P, Ostrowski J, Eatock M, Scheithauer W, Herrmann R, Neoptolemos JP. Phase III randomized comparison of gemcitabine versus gemcitabine plus capecitabine in patients with advanced pancreatic cancer. J Clin Oncol. 2009 Nov 20;27(33):5513-8. doi: 10.1200/JCO.2009.24.2446. Epub 2009 Oct 26. PMID 19858379